CLINICAL TRIAL: NCT00498134
Title: Chemoprevention of Gastric Cancer by Intervention With Helicobacter Pylori and Cyclooxygenase Pathway
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EC1721-01; HARECCTR0500053
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Stomach Neoplasms
Keywords: Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cyclooxygenase 2 Inhibitors

INTERVENTIONS:
Drug: Triple therapy for H. pylori infection
Drug: Cox-2 inhibitor

SUMMARY:
Gastric cancer is the second leading cause of cancer deaths in the World. In China, gastric cancer exceeds all other cancer mortality except lung cancer. Helicobacter pylori infection is an important cause of gastric cancer. We have previously started a randomized placebo-controlled chemoprevention trial in Changle in 1994 to address the issue of whether eradication of H. pylori alone is able to prevent or reduce the risk of gastric cancer. The project involved 1600 subjects and is still ongoing. On the other hand, our laboratory research indicated that an abnormally high expression of an enzyme cyclooxygenase-2 was found in gastric cancer and inhibition of this enzyme by a new drug (specific cyclooxygenase-2 inhibitor) could kill the cancer cells. The same drug is approved now for use in treatment of hereditary colon cancer syndrome (Familial Adenomatous Polyposis, FAP), in the same rationale of tumour suppressive property of this drug. We are now initiating a second chemoprevention study to assess the addition of this specific cyclooxygenase-2 inhibitor together with eradication of H. pylori on prevention or reduction of the risk of gastric cancer and to assess whether the combination can reverse pre-cancerous lesions in the stomach in the high-risk population. The proposed site is Shangdong, China with very high prevalence of pre-cancerous lesions in asymptomatic H. pylori carriers. We plan to recruit 1500 H. pylori positive subjects for this randomized placebo-controlled study. H. pylori carriers will be randomized to receive treatment for the infection or placebo, followed by specific COX-2 inhibitor or placebo for 3 years. The results will have significant impact on prevention of gastric cancer on a national scale and worldwide.

ELIGIBILITY:
Inclusion Criteria:

1. Subject demonstrates a willingness to participate in the study as indicated by written informed consent.
2. Male or female subject is at least 45 years of age.
3. Subject indicates a willingness to abstain from the use of all NSAIDs (including over-the-counter products) and aspirin for the duration of the study.
4. Female subject of childbearing potential has been using an effective means of contraception for 1 week prior to the preliminary visit. She also has agreed to remain abstinent, or to use oral birth control pills or single-barrier contraception (partner using condom or subject using diaphragm, contraceptive sponge or IUD) beginning at the preliminary visit and continuing till the end of the study. Women who are postmenopausal or status post-hysterectomy or tubal ligation are exempt from this requirement. (Postmenopausal is defined as no menses for the previous 1 year. If cessation of menses is within 18 months, FSH must be documented as elevated into the postmenopausal range before entry).
5. Subject is judged to be in stable health based on medical history, physical examination, and routine laboratory tests.

Exclusion Criteria:

According to medical history

1. Subject has a bleeding diathesis or requires anticoagulant therapy.
2. Subject has uncontrolled hypertension. (Note: Subjects with medically controlled hypertension [diastolic blood pressure <95 mm Hg, systolic blood pressure <165 mm Hg] may participate.)
3. Subject has a history of stroke or transient ischemic attack within the past 2 years.
4. Subject has a history of hepatitis/hepatic disease that has been active within the previous 2 years.
5. Subject has angina or congestive heart failure, with symptoms that occur at rest or minimal activity, or has a history of myocardial infarction within the past 1 year.
6. Subject has a history of neoplastic disease within the previous 10 years. Exceptions: subjects with malignancy successfully treated >10 years prior to screening, where, in the judgment of the investigator and treating physician, there has been no evidence of recurrence from the time of treatment through the time of screening.
7. Subject has a history of esophageal or gastric surgery.
8. Subject has undergone previous small or large bowel resection.
9. Subject has a history of inflammatory bowel disease (ulcerative colitis or Crohn's disease).
10. Subject is allergic to paracetamol or subject has hypersensitivity (e.g., all or part of the syndrome of nasal polyps, angioedema, and bronchospastic reactivity) to aspirin, paracetamol, or other NSAIDs. NOTE: Subjects with a history of idiosyncratic allergic reaction (e.g., rash) to a single NSAID in the past but who tolerated at least 2 other NSAID medications without hypersensitivity reactions may participate.
11. Subject is expected to need chronic NSAID treatment during the trial and/or subject has been taking NSAIDs (including salicylates or other aspirin-containing compounds) on a chronic basis.
12. Subject has had ongoing or is expected to require treatment with any of the following: Ticlopidine, clopidrogel, or regular doses of aspirin, including "low-dose" aspirin, e.g., to prevent complications of vascular disease. Subjects may not discontinue an established course of anti-platelet therapy in order to enter this study.

Min Age: 45 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2004-03; Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Regression or prevent progression of various precancerous gastric conditions including gastric atrophy, intestinal metaplasia and dysplasia | 3 years
Changes in cell proliferation, apoptosis and oncogene expressions | 3 years

SECONDARY OUTCOMES:
The incidence of gastric cancer in a high risk area | 5-10 years

CONTACTS AND LOCATIONS:
Overall Officials: Shiu Kum Lam, Prof, Principal Investigator — Department of Medicine, Queen Mary Hospital/ The University of Hong Kong
Locations (1):
- China, China, China